CLINICAL TRIAL: NCT02842372
Title: Non-interventional Study to Investigate Treatment Responses to Topical Application With Ectoin Dermatitis Cream 7% as First-line Therapy of Acute Skin GvHD
Brief Title: Ectoin Dermatitis Cream 7% as First-line Therapy of Acute Skin Graft Versus Host Disease
Status: Withdrawn | Type: Observational
Why Stopped: Study withdrawn due to difficulties in recruiting patients
Sponsor: Bitop AG (Industry)
Responsible Party: Sponsor
Other Study IDs: 2016/EHK02/NIS
Record Dates: First submitted 2016-06-22; First posted 2016-07-22 (Estimated); Last update posted 2018-12-10 (Actual); Status verified 2018-12

CONDITIONS: Acute Graft Versus Host Disease in Skin
Keywords: Acute Graft Versus Host Disease in Skin; GvHD; Ectoin; Dermatitis; Inflammation of the skin; Topical therapy skin GvHD
MeSH Terms: conditions — Dermatitis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Ectoin Dermatitis Cream 7%: Cream for symptomatic treatment and relief of skin redness and itching experienced with various types of inflammatory dermatoses.

SUMMARY:
This is a non-interventional prospective study to investigate the treatment response to topical application with Ectoin Dermatitis Cream 7% as first-line therapy of grade I acute skin graft-versus-host disease.

DETAILED DESCRIPTION:
Graft-versus-host disease (GvHD) is a medical complication following the receipt of transplanted tissue from a genetically different person. In the classical sense, acute graft-versus-host-disease is characterized by selective damage to different organ systems and the severity of acute GVHD is determined by an assessment of the degree of involvement of the skin, liver, and gastrointestinal tract.

In general topical steroids can be used as first line treatment in acute grade I skin GvHD according to Dignan et al 2012. However, the administration of high doses and/or prolonged use of topical steroids is associated with severe side effects, such as opportunistic infections, that is a significant factor for morbidity and mortality. Furthermore, the results of corticosteroid treatment are clearly suboptimal, with continuing complete response rates of only 20-40% in acute and chronic GVHD. Therefore, it still remains a matter of debate whether there is an alternative first line therapy to topical steroids that can overcome these problems.

Ectoin Dermatitis Cream is a high quality cream containing 7% Ectoin without cortisone for the symptomatic, proactive treatment of atopic dermatitis or other inflammatory skin diseases as e.g. radio or contact dermatitis. In several clinical studies it has been shown that Ectoin Dermatitis Cream reduces inflammation of the skin during sub-acute periods and stabilizes the skin barrier. In acute periods, it reduces the symptoms like itchiness and redness of the skin.

In this study, Ectoin Dermatitis Cream can be used as therapy of grade 1 (stage 1 and 2) acute skin GvHD in patients who have a hypersensitivity to corticosteroids or show an ineffectiveness of topical corticosteroids. Following confirmation of the diagnosis, patients will asked by the investigator whether they are interested to participate in the current trial. The investigator, taking the patients into consideration is free to decide who is to receive the Ectoin Dermatitis Cream.

Patients enrolled in this observational trial will be treated for 14 days with Ectoin Dermatitis Cream. Patients who do not respond to Ectoin therapy within the first 5 to 7 days of treatment, will be treated with topical or systemic steroids. However, when there are indications of good treatment response, the patients will be treated with Ectoin Dermatitis Cream until symptoms resolve.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of acute skin graft versus host disease grade I
* hypersensitivity to corticosteroids or ineffectiveness of topical corticosteroids

Exclusion Criteria:

* Grade II-IV GVHD (history of or at time of study entry)
* Use of any systemic steroids at any time for GVHD Treatment
* Non-compliance with medication
* Allergic or otherwise undesirable reaction to Ectoin or any of the other ingredients of the topical cream
* Patients with exanthema of the face
* Pre-existing dermatologic conditions (e.g. eczema, psoriasis, acne etc.)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with acute skin GvHD grade I (stage 1 or 2) who have either a hypersensitivity to corticosteroids or who are characterized by an ineffectiveness of topical corticosteroids.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2015-12; Primary Completion 2018-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Change in severity of skin GvHD as assessed by a visual examination and asking the patient about pain and discomfort | Visit 1 (day 0), Visit 2 (after 7±2 days), Visit 3 (after 14±2 days)
  A trained clinical member of the team scores the degree and severity of skin GvHD as follow: stage 1, maculopapular rash over <25 percent of body area; stage 2, maculopapular rash over 25 to 50 percent of body area; stage 3, generalized erythroderma; stage 4, generalized erythroderma with bullous formation, often with desquamation
The number of patients who progress within 14 days of initiation of Ectoin treatment | 14 days after starting treatment with Ectoin Dermatitis Cream
Change in intensity of itching by using a patient-reported experience questionnaire | Visit 1 (day 0), Visit 2 (after 7±2 days), Visit 3 (after 14±2 days)
  The intensity of itching will be graded on a numeric scale, i.e. absent-0, severe-10
Change in Evaluation of touch sensitivity by using a patient-reported experience questionnaire | Visit 1 (day 0), Visit 2 (after 7±2 days), Visit 3 (after 14±2 days)
  The intensity of touch sensitivity will be graded on a numeric scale, i.e. absent-0, severe-10
Change in Evaluation of limited mobility by using a patient-reported experience questionnaire | Visit 1 (day 0), Visit 2 (after 7±2 days), Visit 3 (after 14±2 days)
  The intensity of limited mobility will be graded on a numeric scale, i.e. absent-0, severe-10
Change in Evaluation of pain by using a patient-reported experience questionnaire | Visit 1 (day 0), Visit 2 (after 7±2 days), Visit 3 (after 14±2 days)
  The intensity of pain will be graded on a numeric scale, i.e. absent-0, severe-10
Change in Evaluation of wounds by using a patient-reported experience questionnaire | Visit 1 (day 0), Visit 2 (after 7±2 days), Visit 3 (after 14±2 days)
  The intensity of wounds will be graded on a numeric scale, i.e. absent-0, severe-10
Change in Evaluation of inflammation of Skin by using a patient-reported experience questionnaire | Visit 1 (day 0), Visit 2 (after 7±2 days), Visit 3 (after 14±2 days)
  The intensity of inflammation will be graded on a numeric scale, i.e. absent-0, severe-10
Change in intensity of erythema evaluated by the physician | Visit 1 (day 0), Visit 2 (after 7±2 days), Visit 3 (after 14±2 days)
  The intensity of erythema will be graded on a 4-point scale, i.e. 0-absent, severe-4
Change in Evaluation of dry Skin evaluated by the physician | Visit 1 (day 0), Visit 2 (after 7±2 days), Visit 3 (after 14±2 days)
  The intensity of dry Skin will be graded on a 4-point scale, i.e. 0-absent, severe-4
Change in Evaluation of hyperkeratosis evaluated by the physician | Visit 1 (day 0), Visit 2 (after 7±2 days), Visit 3 (after 14±2 days)
  The intensity will be graded on a 4-point scale, i.e. 0-absent, severe-4
Change in Evaluation of rhagades evaluated by the physician | Visit 1 (day 0), Visit 2 (after 7±2 days), Visit 3 (after 14±2 days)
  The intensity will be graded on a 4-point scale, i.e. 0-absent, severe-4

SECONDARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | within 14 days after starting treatment with Ectoin Dermatitis Cream

CONTACTS AND LOCATIONS:
Overall Officials: Martina Haibach, PhD, Principal Investigator — Universitätsklinikum Erlangen
Locations (1):
- Department of medicine 5, Haematology and Oncology, University hospital Erlangen, Erlangen, Germany

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Dignan FL, Clark A, Amrolia P, Cornish J, Jackson G, Mahendra P, Scarisbrick JJ, Taylor PC, Hadzic N, Shaw BE, Potter MN; Haemato-oncology Task Force of British Committee for Standards in Haematology; British Society for Blood and Marrow Transplantation. Diagnosis and management of acute graft-versus-host disease. Br J Haematol. 2012 Jul;158(1):30-45. doi: 10.1111/j.1365-2141.2012.09129.x. Epub 2012 Apr 26. PMID 22533831